CLINICAL TRIAL: NCT01844570
Title: Levamlodipine Maleate (Xuanning) or Amlodipine Besylate (Norvasc) for Treatment of Hypertension: A Comparative Effectiveness Research
Brief Title: Levamlodipine Maleate or Amlodipine Besylate for Treatment of Hypertension: A Comparative Effectiveness Research
Acronym: LEADER
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Peking University First Hospital (Other)
Collaborators: Ministry of Science and Technology of the People´s Republic of China (Other Government); Southern Medical University, China (Other); CSPC Ouyi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Yong Huo, Professor of cardiovascular medicine, Peking University First Hospital
Other Study IDs: LEADER
Record Dates: First submitted 2013-04-28; First posted 2013-05-01 (Estimated); Last update posted 2013-05-01 (Estimated); Status verified 2013-04

CONDITIONS: Primary Hypertension
MeSH Terms: conditions — Essential Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Levamlodipine Maleate (Xuanning): Primary hypertensive patients who take Levamlodipine Maleate (Xuanning) as the only anti-hypertensive medication or one of their medications
- Amlodipine Besylate (Norvasc): Primary hypertensive patients who take Amlodipine Besylate (Norvasc) as the only anti-hypertensive medication or one of their medications

SUMMARY:
The purpose of this study is to determine whether the effectiveness of levamlodipine maleate (xuanning) is noninferior to amlodipine besylate (Norvasc) in treatment of hypertension in a Chinese primary hypertension population.

DETAILED DESCRIPTION:
It is a multicenter, prospective cohort study with large sample size. It is to evaluate the effect on the incidence of cardiovascular and cerebrovascular endpoint events and blood pressure control in hypertensive patients who use Levamlodipine Maleate (Xuanning) or amlodipine besylate(Norvasc).Xuanning group and Norvasc group will recruit 5000 patients respectively. Each site will recruit patients in chronological order；patients who participate will finish the two-year follow up(1,2,3,6,12,18,24 months after recruitment) and relevant data will be recorded. Baseline data will be analyzed to evaluate the equilibrium between two or more groups (such as the number of options). Logistic regression and propensity scores (PS) would be used to match major indicators of effectiveness and safety indicators using matching method baseline data.

ELIGIBILITY:
Inclusion Criteria:

* systolic pressure ≥140mmHg or diastolic pressure ≥90mmHg or receiving antihypertensive drug treatment
* Patient himself/herself or his/her family member has already signed the informed consent form
* Patient is fit for use of Levamlodipine Maleate or amlodipine besylate
* Age≥45

Exclusion Criteria:

* patient with secondary hypertension
* patients who has suffered from myocardial infarction or stroke within the latest 3 months
* patients who has obvious intelligence、hearing and limb's activity disability
* Patients with severe disease, with a life expectancy of less than two years

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 eligible sites(including primary care clinic and tertiary hospitals) over the country will participate. Each center will collect patients who fit the recruitment standard in chronological order.
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2013-02; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
incidence of composite cardiovascular and cerebrovascular endpoints | 2 years
quality of blood pressure control | 2 years

SECONDARY OUTCOMES:
incidence of adverse reaction | 2 years
cost-effectiveness analysis | 2 years
Explore the optimal combination of drugs for the treatment of hypertension by Levamlodipine Maleate | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Yong Huo, MD, Principal Investigator — Department of Cardiology, Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, China

REFERENCES:
- [Derived] Ma W, Sun N, Duan C, Zhao L, Hua Q, Sun Y, Dang A, Gao P, Qu P, Cui W, Zhao L, Dong Y, Cui L, Qi X, Jiang Y, Xie J, Li J, Wu G, Du X, Huo Y, Chen P; for LEADER Study Group. Effectiveness of Levoamlodipine Maleate for Hypertension Compared with Amlodipine Besylate: a Pragmatic Comparative Effectiveness Study. Cardiovasc Drugs Ther. 2021 Feb;35(1):41-50. doi: 10.1007/s10557-020-07054-1. Epub 2020 Sep 11. PMID 32915349